CLINICAL TRIAL: NCT02543684
Title: Post-prandial Glucose and Insulin Levels in Type 2 Diabetes Mellitus Patients After Consumption of Ready-to-eat Mixed Meals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harokopio University (Other)
Responsible Party: Principal Investigator, Yannis Manios, Associate Professor, Harokopio University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Diabetes study
Record Dates: First submitted 2015-09-03; First posted 2015-09-07 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: glycemic response; diabetes; insulinemic response; mixed meals; glycemic index
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

ARMS (4):
- ready to eat mixed meal 1 (Experimental)
  Interventions: Other: ready to eat mixed meal 1
- ready to eat mixed meal 2 (Experimental)
  Interventions: Other: ready to eat mixed meal 2
- ready to eat mixed meal 3 (Experimental)
  Interventions: Other: ready to eat mixed meal 3
- oral glucose load (Experimental)
  Interventions: Other: oral glucose load

INTERVENTIONS:
Other: ready to eat mixed meal 1 — wild greens pie providing 50g of carbohydrates
  Other Names: Sunday's Catering Company
  Arms: ready to eat mixed meal 1
Other: ready to eat mixed meal 2 — chicken burgers with boiled broccoli and cauliflower providing 50g of carbohydrates
  Other Names: Sunday's Catering Company
  Arms: ready to eat mixed meal 2
Other: ready to eat mixed meal 3 — vegetable moussaka providing 50g of carbohydrates
  Other Names: Sunday's Catering Company
  Arms: ready to eat mixed meal 3
Other: oral glucose load — glucose load providing 50g of carbohydrates
  Arms: oral glucose load

SUMMARY:
The aim of the current study was to compare the effects of three ready-to-eat mixed meals, with a high fiber content and low glycemic index, on postprandial glycemic and insulinemic response in patients with Type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
The current study followed a prospective, three-way, cross-over design. Twenty four patients with T2DM consumed three ready-to-eat mixed meals, i.e. "wild greens pie" (meal 1), "chicken burgers with boiled vegetables" (meal 2) and "vegetable moussaka" (meal 3) and an oral glucose load, all providing 50g of carbohydrates. Venous blood was collected at 0, 30, 60, 90 and 120 minutes postprandial for serum glucose and insulin measurements.

The test meals were consumed by study participants between 8:30 to 9:00 am and within 10-15 minutes under a researcher's supervision, following collection of the fasting blood sample. No parallel fluid intake was allowed. The portion size in the case of each one of the three test meals was adjusted to contain 50g of carbohydrates. However, the three test meals were considerably differentiating among them with respect to their content in calories and the remaining macronutrients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are eligible if they are 45-75 years of age
* non-insulin-dependent T2DM with an elapsed time since diagnosis of more than 3 years
* Body Mass Index (BMI) value higher than 20 kg/m2
* HbA1c levels of 6.5 to 11%

Exclusion Criteria:

* insulin-dependent T2DM
* cardiovascular (i.e. coronary heart disease, stroke etc.)
* liver and/or renal disease

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-11; Primary Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
serum glucose changes over time | fasting baseline glucose at time 0, then 30, 60, 90, and 120 minutes postprandial
serum insulin changes over time | fasting baseline insulin at time 0, then 30, 60, 90, and 120 minutes postprandial

CONTACTS AND LOCATIONS:
Overall Officials: Yannis Manios, Associate Professor, Principal Investigator — Harokopio University, Athens
Locations (1):
- Harokopio University of Athens, Kallithea, Attica, Greece